CLINICAL TRIAL: NCT05916417
Title: TMS-fNIRS Personalized Dosing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, F. Andrew Kozel, Professor & Mina Jo Powell Endowed Chair, Neurological Sciences, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00004007; CDMRP-TP220192 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-05-15; First posted 2023-06-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Post Traumatic Stress Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: A total of 60 participants will be recruited and assigned to one of the two arms (active or sham TMS) at a 4:1 ratio (i.e., 48 participants for the active TMS group and 12 for the sham group).
  The primary outcome is the MC or dl-PFC fNIRS signal, and a total of 12 comparisons will be conducted (i.e., one test for Aim 1; one for Aim 2; and 10 for Aim 3, considering the comparisons of CNR and TDR for the four longer paradigms as well as the shorter paradigm).
Who Masked: Participant, Investigator
Masking Description: Blinding Procedures The participants, PI, Research Staff involved in TMS treatment, and staff performing the study procedures will be blinded to the participant's dl-PFC protocol assignment throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- TMS-fNIRS over the dl-PFC (Active) (Active Comparator): TMS-fNIRS dl-PFC data will be acquired with participants being randomized to active or sham stimulation of the dl-PFC, with the randomizing of the order of four different TMS-fNIRS protocols.
  Interventions: Device: TMS-fNIRS over the dl-PFC
- TMS-fNIRS over the dl-PFC (Sham) (Sham Comparator): TMS-fNIRS dl-PFC data will be acquired with participants being randomized to active or sham stimulation of the dl-PFC, with the randomizing of the order of four different TMS-fNIRS protocols.
  Interventions: Device: TMS-fNIRS over the dl-PFC

INTERVENTIONS:
Device: TMS-fNIRS over the dl-PFC — Transcranial Magnetic Stimulation (TMS) is a non-invasive brain stimulation technology. Functional Near Infrared Spectroscopy (fNIRS) is a brain imaging technology that utilizes light.

SUMMARY:
The intent of this study is to establish technical feasibility in a clinical population (PTSD, with or without mild TBI) of personalized TMS-fNIRS technology. Thereby demonstrating the utility of transcranial magnetic stimulation - functional near-infrared spectroscopy (TMS-fNIRS) technology as a direct measure of frontal brain activity, potentially replacing the indirect motor threshold procedure that may lead to improper dosing of TMS.

Personalized TMS-fNIRS technology will guide therapy for depression, post-traumatic stress disorder (PTSD), and/or traumatic brain injury (TBI)

ELIGIBILITY:
Inclusion Criteria

1. Adults ages 18-70 years.
2. Eligible for consideration of treatment with TMS for PTSD.
3. Diagnosis of PTSD based on CAPS-5.
4. No changes in psychotropic medication (if taking psychotropic medication) and/or changes in supportive psychotherapy for 1 month prior to initial visit; and clinically appropriate to maintain stable treatment regimen for duration of study.
5. Clinically competent to give informed written consent and ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

1. Medical contraindication for neuromodulation (e.g., ferrous metal in head, seizure disorder, brain tumor, stroke, aneurysm, multiple sclerosis, etc.).
2. Unable to have an MRI (e.g., due to ferrous metal or inability to tolerate).
3. Active substance use disorder in last 3 months or any current substance use that puts the participant at increased risk or significant impairment
4. Dementia or other cognitive disorder making unable to engage in study.
5. Any history or diagnosis of Schizophrenia, Schizoaffective Disorder, Delusional Disorder or other psychotic illness.
6. Suicidal risk that precludes safe participation defined as clinical impression that the participant is at significant risk for suicide.
7. OCD cannot be the primary disorder but can have OCD symptoms
8. Taking any medication that significantly lowers the seizure threshold (e.g., tricyclic antidepressants, clozapine, etc.)
9. Current, planned, or suspected pregnancy
10. Unstable medical conditions or any current medical condition that could preclude being able to safely participate in TMS treatment (e.g., unstable metabolic abnormality, unstable angina, etc.)
11. Severe Traumatic Brain Injury
12. Prior TMS treatment or already received TMS as part of a study.
13. Significant ongoing litigation or claims that impact research activities, as determined by the research study team. (Research may especially be impacted when mental health or pain is being evaluated for litigation or claims, such as civil and criminal cases, disability claims and worker's compensation).

We will exclude non-English speakers because of the need for rapid communication during the testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
TMS induced Brain changes as measured by functional Near Infrared Spectroscopy (fNIRS) comparing Motor Cortex (MC) and Dorsolateral Prefrontal Cortex (dl-PFC) | Months 3-33
  The magnitude of brain activation based on fNIRS signal for the respective cortices at the individual level will be assessed and compared for the MC and dl-PFC.

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Kozel, M.D., M.S.C.R., D.F.A.P.A., Principal Investigator — Florida State University
Locations (1):
- Isabelle Taylor, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT05916417/ICF_000.pdf